CLINICAL TRIAL: NCT02353689
Title: Identification of the Effect of Fermentable Oligo-, di-, and Mono- Saccharides and Poorly Absorbed Short-chain Carbohydrate (FODMAP) Content in Tube Feeding Formula on Feeding Intolerance and Nutritional Status Improvement
Brief Title: The Effect of FODMAP Content in Tube Feeding Formula on Feeding Intolerance and Nutritional Status Improvement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oh Yoen Kim (Other)
Collaborators: Dong-A University (Other)
Responsible Party: Sponsor-Investigator, Oh Yoen Kim, Assistant Professor, Dong-A University
Organization: Dong-A University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2-1040709-AB-N-01-201310-BR-03
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Enteral Nutrition
MeSH Terms: interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low FODMAP group (Experimental): consumed EN formula containing low FODMAPs (0.320g/can) during 14-day intervention
  Interventions: Dietary Supplement: low FODMAP
- moderate FODMAP group (Experimental): consumed EN formula containing moderate FODMAPs (0.753g/can) during 14-day intervention
  Interventions: Dietary Supplement: moderate FODMAP
- high FODMAP group (Experimental): consumed EN formula containing high FODMAPs (1.222g/can) during 14-day intervention
  Interventions: Dietary Supplement: high FODMAP

INTERVENTIONS:
Dietary Supplement: low FODMAP — consumed EN formula containing low FODMAPs (0.320g/can) during 14-day intervention
  Arms: low FODMAP group
Dietary Supplement: moderate FODMAP — consumed EN formula containing moderate FODMAPs (0.753g/can) during 14-day intervention
  Arms: moderate FODMAP group
Dietary Supplement: high FODMAP — consumed EN formula containing high FODMAPs (1.222g/can) during 14-day intervention
  Arms: high FODMAP group

SUMMARY:
This study aimed to investigate the effects of FODMAP contents in enteral nutrition (EN) formulas on major gastrointestinal intolerance symptoms and nutritional status in tube fed patients through the randomized, double blind and placebo-controlled trial.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on 100 tube-fed patients. Over a 14-day test period, the test group consumed EN formula containing low FODMAPs, while the placebo groups consumed EN formula containing moderate or high FODMAPs .

ELIGIBILITY:
Inclusion Criteria:

* tube-feeding patients

Exclusion Criteria:

* EN prohibited
* renal dysfunction (i.e. serum creatinine > 1.5 mg/dl or blood urea nitrogen > 25 mg/ml)
* liver dysfunction (i.e. serum aspartate aminotransferase > 40 U/L or alanine aminotransferase > 40 U/L)
* uncontrollable diabetes mellitus
* pregnancy, breast-feeding etc.
* severe diarrhea

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
diarrhea | 14-day follow-up

SECONDARY OUTCOMES:
prealbumin | 14-day follow-up
body mass index | 14-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Oh Yoen Kim, PhD, Principal Investigator — Dong-A Univeristy